CLINICAL TRIAL: NCT05067309
Title: Termination of Early Pregnancy in Scarred Uterus With Letrozole and Misoprostol Compared to Misoprostol Alone
Brief Title: Termination of Early Pregnancy in Scarred Uterus With Lletrozole and Misoprostol Compared to Misoprostol Alone
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Elsayed Aref (Other)
Responsible Party: Sponsor-Investigator, Ahmed Elsayed Aref, Ahmed Elsayed Aref, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-21-09-07
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Termination of Early Pregnancy in Scarred Uterus
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Missed abortion received letrozole then misoprostol
  Interventions: Drug: Letrozole 2.5mg
- Missed abortion received misoprostol alone

INTERVENTIONS:
Drug: Letrozole 2.5mg — Missed abortion received letrozole then misoprostol
  Groups: Missed abortion received letrozole then misoprostol

SUMMARY:
Termination of early pregnancy in scarred uterus with letrozole and misoprostol compared to Misoprostol alone

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years for mother.

  * Non-viable fetus (missed abortion or blighted ovum) in the 1st trimester of pregnancy evidenced by criteria for diagnosis by TVS .
  * Previous C.S or Myomectomy (1 or more )
  * lack of any maternal diseases such as: heart disease, asthma, history of thromboembolism, cancer, renal failure, and liver diseases.

Exclusion Criteria:

* * Medical problem in patient

  * Emergency conditions which need intervention .
  * History of allergy to misoprostol or letrozole drugs.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Termination of early pregnancy in scarred uterus with letrozole and misoprostol compared to Misoprostol alone
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete abortion of early pregnancy with letrozole then misoprostol | 6 months
  Letrozole increase cervical ripening

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Elsayed Aref, Sohag, Egypt